CLINICAL TRIAL: NCT06914791
Title: Differential Rehabilitative Treatment for Pelvic Floor in Sportswoman: an Interventional Pilto Study Comparing Kegel and De Gasquet Approach
Brief Title: Differential Rehabilitative Treatment for Pelvic Floor in Sportswoman
Acronym: DiRehFloor
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alessandro Micarelli (Other)
Responsible Party: Sponsor-Investigator, Alessandro Micarelli, Scientific Director - Principal Investigator, Uniter Onlus
Organization: Uniter Onlus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PelvicRehab1
Record Dates: First submitted 2025-03-22; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Floor Disorder
Keywords: pelvic floor rehabilitation
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kegel arm (Active Comparator)
  Interventions: Procedure: Kegel arm
- De Gasquet arm (Experimental)
  Interventions: Procedure: De Gasquet arm

INTERVENTIONS:
Procedure: Kegel arm — in this group participants will be followed up for 8 weeks with kegel exercises
  Arms: kegel arm
Procedure: De Gasquet arm — in this group participants will be followed up for 8 weeks with de gasquet exercises
  Arms: De Gasquet arm

SUMMARY:
In this study at least 24 sportswoman (18-50 years old) will be recruited a randomized in two groups which will be differently treated for the following 8 weeks. one group will be treated with Kegel approach and the other one with De Gasquet apporach. before and after the treatment they will fill in a battery of falidated questionnaire in order to evaluate the improvement at pelvic floor level, quality of life and psychological distress.

DETAILED DESCRIPTION:
In this study at least 24 sportswoman (18-50 years old) with pelvic floow symptos (18-50 years old) will be recruited a randomized in two groups which will be differently treated for the following 8 weeks. They should havo no children, other relevant systemic disorders and assume no drugs. They should practice sports by at least one year.

one group will be treated with Kegel approach and the other one with De Gasquet apporach. before and after the treatment they will fill in a battery of falidated questionnaire in order to evaluate the improvement at pelvic floor level, quality of life and psychological distress. In partiqular they fill in:

* Pelvic Floor Distress Inventory (PFDI-20)
* Incontinence Severity Index (ISI)
* Quality of life questionnaire (SF-36)
* King's Health Questionnaire (KHQ)
* Intestinal related symptoms questionnaire (ICIQ-B)
* Depression Anxiety Stress Scale (DASS-21)

ELIGIBILITY:
Inclusion Criteria:

* practicing sports by at least one year

Exclusion Criteria:

* no systemic disorders
* no drugs assumption
* no children

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory (PFDI-20) | 8 weeks
  Pelvic Floor Distress Inventory evalueates the pelvic floor distress with values ranging from 0 to 300 indicating respectively better and worse score

SECONDARY OUTCOMES:
Incontinence Severity Index (ISI) | 8 weeks
  the Incontinence Severity Index evaluates the incontinence with values ranging from 0 to 12 indicating respectively better and worse score
Quality of life questionnaire (SF-36) | 8 weeks
  the Quality of life questionnaire evaluates the quality of life with values ranging from 0 % to 100 % indicating respectively better and worse limitations
King's Health Questionnaire (KHQ) | 8 weeks
  the King's Health Questionnaire evaluates the urinary tract consequences on daily life with values ranging from 0 to 100 indicating respectively better and worse limitations
Intestinal related symptoms questionnaire (ICIQ-B) | 8 weeks
  the Intestinal related symptoms questionnaire evaluates the intestinal consequences on daily quality of life with values ranging from 0 to 26 indicating respectively better and worse scores
Depression Anxiety Stress Scale (DASS-21) | 8 weeks
  Depression Anxiety Stress Scale evaluates anxiety, depression and stress with values ranging from 0 to 14 indicating respectively better and worse scores for depression, 0 to 10 indicating respectively better and worse scores for anxiety and 0 to 17 indicating respectively better and worse scores for stress

CONTACTS AND LOCATIONS:
Locations (1):
- UNITER Onlus Foundation, Fara in Sabina, Italy

IPD SHARING:
Plan to Share IPD: No
it is not possible for the law of our contry

REFERENCES:
- [Result] Campbell KG, Batt ME, Drummond A. Prevalence of pelvic floor dysfunction in recreational athletes: a cross-sectional survey. Int Urogynecol J. 2023 Oct;34(10):2429-2437. doi: 10.1007/s00192-023-05548-8. Epub 2023 May 10. PMID 37162534
- [Result] Brandt F, Solomayer EF, Sklavounos P. Correlation between the Incontinence Severity Index (ISI) and the quality of life dimensions of the King's Health Questionnaire (KHQ) in German-speaking urinary incontinent women. J Gynecol Obstet Hum Reprod. 2022 Feb;51(2):102288. doi: 10.1016/j.jogoh.2021.102288. Epub 2021 Dec 10. PMID 34902634
- [Result] Bø K. Exercise and Pelvic Floor Dysfunction in Female Elite Athletes. Handbook of Sports Medicine and Science: The Female Athlete. 2015
- [Result] Blazek D, Stastny P, Maszczyk A, Krawczyk M, Matykiewicz P, Petr M. Systematic review of intra-abdominal and intrathoracic pressures initiated by the Valsalva manoeuvre during high-intensity resistance exercises. Biol Sport. 2019 Dec;36(4):373-386. doi: 10.5114/biolsport.2019.88759. Epub 2019 Oct 17. PMID 31938009
- [Result] Barba M, Cola A, Melocchi T, Braga A, Castronovo F, Manodoro S, Pennacchio M, Munno GM, Ruffolo AF, Degliuomini RS, Salvatore S, Torella M, Frigerio M. Italian validation of the Pelvic Floor Distress Inventory (PFDI-20) questionnaire. Int Urogynecol J. 2023 Oct;34(10):2459-2465. doi: 10.1007/s00192-023-05572-8. Epub 2023 May 17. PMID 37195425
- [Result] Alves JO, Luz STD, Brandao S, Da Luz CM, Jorge RN, Da Roza T. Urinary Incontinence in Physically Active Young Women: Prevalence and Related Factors. Int J Sports Med. 2017 Nov;38(12):937-941. doi: 10.1055/s-0043-115736. Epub 2017 Sep 26. PMID 28950397
- [Result] Almeida MB, Barra AA, Saltiel F, Silva-Filho AL, Fonseca AM, Figueiredo EM. Urinary incontinence and other pelvic floor dysfunctions in female athletes in Brazil: A cross-sectional study. Scand J Med Sci Sports. 2016 Sep;26(9):1109-16. doi: 10.1111/sms.12546. Epub 2015 Sep 15. PMID 26369504
- [Result] Abd El-Aty E.M., Hassan M.E.-G. Effect of Kegel Exercise Training Program On Improving Quality Of Life Among Women With Urinary Incontinence. Egypt. J. Health Care. 2021